CLINICAL TRIAL: NCT04793438
Title: Treating Negative Symptoms of Schizophrenia With a Motive-specific Intervention: A Randomised Controlled Trial
Brief Title: Motive-specific Intervention for Negative Symptoms in Schizophrenia
Acronym: MoNSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-00916
Record Dates: First submitted 2018-09-06; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Negative Type; Schizophrenic; Anhedonia; Apathy
Keywords: Negative symptoms; Psychosis; Schizophrenia; Psychotherapy; Inpatients; Apathy; Anhedonia; Avolition
MeSH Terms: conditions — Anhedonia; Lethargy; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Motive-specific intervention; three appointments within two weeks, 30-45 minutes per session.
  Interventions: Behavioral: Motive-specific intervention
- Control group (Active Comparator): Supportive conversations; three appointments within two weeks; 30-45 minutes per session.
  Interventions: Behavioral: Supportive conversations

INTERVENTIONS:
Behavioral: Motive-specific intervention — Three appointments are made with the patients of the intervention group within two weeks. With an adaptation of the Autobiographical Memory Test (AMT) participants will be asked to recall events from the past and to imagine future events. The time frame of 45 minutes for each intervention must be strictly adhered to. Patients are additionally asked to complete tasks between the sessions. All appointments take place in the Psychiatric University Hospital directly on the ward.
  Arms: Intervention group
Behavioral: Supportive conversations — Since we want to check whether the patients benefit from the specific intervention and not only from getting more speaking time, patients without the motive-specific intervention should also be given three sessions, in which no intervention takes place. They will be carried out in the sense of supportive conversations (i.e. conversations that do not follow a specific psychotherapy concept). All appointments take place in the Psychiatric University Hospital directly on the ward.
  Arms: Control group

SUMMARY:
The aim of this study is to test a therapeutic intervention to reduce negative symptomatic among schizophrenia patients. Since the intervention can take place within an inpatient stay, it is a short intervention. Three appointments are made with the patients within two weeks. With an adaptation of the Autobiographical Memory Test (AMT) participants will be asked to recall events from the past and to imagine future events. Patients are additionally asked to complete tasks between the sessions. One pre- and one post-measurement of negative symptoms, motives, level of functioning, hope for recovery and other co-variables are part of the study. A follow-up appointment four weeks later is intended to provide information on the longer-term impact.

DETAILED DESCRIPTION:
Clinically relevant negative symptoms are present in almost 60% of all patients suffering from schizophrenia. Motivational deficits seem to be one of the main barriers in the process of "functional recovery" among those patients and have been shown to be very treatment resistant. Effects of pharmacological compounds are at best moderate. There are some psychotherapeutic intervention studies that show promise but further controlled trials are needed to clarify the specific treatment effects.

Therefore, patients shall be encouraged to remember memories that stand in an association with specific motives. Motives are conscious and unconscious affect-based needs that are activated by behavior and influence behavior toward specific incentives in specific circumstances. They influence the selection of everyday goals and have influence on the degree of the progress people are making towards these goals. The intervention is based on the assumption that a positive expectation of the future is constituted among others by positive experiences from the past and at the same time increases the motivation for future behaviour. The activation of specific, motive-associated memories from autobiographical memory and their transformation into images of the future by means of imaginative methods could be a possible way of strengthening certain motives and thus increasing motivation for certain behaviour. This is mainly because there is evidence that psychosis patients have difficulties specifically remembering memories, i.e. those that happened on only one day. In addition, there is a diminished ability to create specific images of their personal future.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male and female inpatients between 18 and 65 years of age
* ICD-10 diagnosis of psychosis (F2)
* Clinical relevant negative symptoms
* Ability to judge with regard to decisions on study participation
* Fluent in German and able to understand the instructions

Exclusion Criteria:

* Florid positive psychotic symptoms (measured with PANSS; that is any positive-subscale item score higher than five)
* Post-schizophrenic depression (ICD: F20.4)
* Organic schizophrenia-like disorder (ICD: F0.6)
* Known or suspected non-compliance, drug or alcohol abuse during treatment
* Cognitive impairments: strongly below average values in cognitive tests
* Complete stop or restart of taking antipsychotic medication during the study (dose adjustments are not a reason for exclusion)
* Previous enrolment in the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of negative symptoms measured with the Brief Negative Symptom Scale (BNSS) | Baseline
  The primary outcome criterion is the change and expected reduction of the severity of the negative symptoms in schizophrenia patients before and after the three-week motive-specific intervention. We compare the change of severity between the patients of the intervention group and those in the control group. Negative symptoms are measured with the Brief Negative Symptom Scale (BNSS) and items are rated on a 7-point-scale (0 = absent, 6 = severe).
Long-term Reduction of negative symptoms measured with the Brief Negative Symptom Scale (BNSS) | 4 weeks after end of the psychotherapeutic intervention
  Another primary outcome criterion is the change of the severity of the negative symptoms in schizophrenia patients who have received the motive-specific intervention compared to the control group patients in a follow-up appointment four weeks after termination of the intervention. Negative symptoms are measured with the Brief Negative Symptom Scale (BNSS) and items are rated on a 7-point-scale (0 = absent, 6 = severe).

SECONDARY OUTCOMES:
Correlation between the severity of negative symptoms and explicit motives measured with the Questionnaire for the Zurich Model of Social Motivation | Baseline
  Secondary outcome criterion is the statistical significance and quality of the relationship between negative symptoms (measured with the Brief Negative Symptom Scale; items are rated on a 7-point-scale with 0 = absent and 6 = severe) and explicit reported motives.
Correlation between the severity of negative symptoms and implicit motives measured with the Multi Motive Gitter | Baseline
  Another secondary outcome criterion is the statistical significance and quality of the relationship between negative symptoms (measured with the Brief Negative Symptom Scale; items are rated on a 7-point-scale with 0 = absent and 6 = severe) and implicit motives.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Kleim, Prof. Dr., Principal Investigator — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No